CLINICAL TRIAL: NCT03570580
Title: Inter Scorers Agreement for OSA Screening Scores.
Status: Completed | Type: Observational
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Head of Department, Astes
Other Study IDs: SEED-COMP
Record Dates: First submitted 2018-06-16; First posted 2018-06-27 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea, Obstructive, Mass Screening
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main Group - OSA Scoring: All patients include in this study for whom the four OSA scoring will be evaluated
  Interventions: Other: OSA scoring

INTERVENTIONS:
Other: OSA scoring — OSA scoring (four scores: STOP-Bang, P-SAP, OSA50, DES-OSA were performed by several scorers on each patients, after what agreement between scores will be evaluated).

SUMMARY:
Four scores are usually performed to detect OSA (Obstructive Sleep Apnea) patients. These four scores are: STOP-Bang, P-SAP, OSA50 and DES-OSA. These scores have been previously validated. However, a comparison between scorers in the realization of these scores has never been performed.

DETAILED DESCRIPTION:
Four scores are usually performed to detect OSA (Obstructive Sleep Apnea) patients. These four scores are: STOP-Bang, P-SAP, OSA50 and DES-OSA. These scores have been previously validated. However, a comparison between scorers in the realization of these scores has never been performed. The aim of this study was to evaluate this agreement using statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* All preoperative patients in the Cabinet Medical ASTES

Exclusion Criteria:

* Patient's refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For all the patients include in the study, the four scores (STOP-Bang, P-SAP, OSA50, and DES-OSA) will be performed several times by various scorers.
  The agreement between scorers will be statistically evaluated.
Sampling Method: Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
OSA Scoring | 2 months
  Should the inter-scorers agreement between OSA scoring be accurate?

CONTACTS AND LOCATIONS:
Overall Officials: Eric Deflandre, MD, PhD, Principal Investigator — Astes
Locations (1):
- Clinique Saint-Luc Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Undecided